CLINICAL TRIAL: NCT03656068
Title: A Monocentric, Open-Label, Proof of Concept Study to Evaluate the Safety and Efficacy of Nitazoxanide at 500mg Twice Daily on Collagen Turnover in Plasma in NASH Patients With Fibrosis Stage 2 or 3
Brief Title: An Evaluation of the Safety and Efficacy of Nitazoxanide on Collagen Turnover in NASH Patients With Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pinnacle Clinical Research, PLLC (Other)
Responsible Party: Principal Investigator, Stephen A. Harrison, Principal Investigator, Pinnacle Clinical Research, PLLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NTZ-218-1
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Non-alcoholic Steatohepatitis; Fatty Liver; Fibrosis, Liver; Compensated Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis | interventions — nitazoxanide; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label NTZ (Experimental): Open label. All patients will receive study drug
  Interventions: Drug: Nitazoxanide 500mg BID

INTERVENTIONS:
Drug: Nitazoxanide 500mg BID — Patients will receive 500mg of Nitazoxanide BID daily for 24 weeks
  Other Names: NTZ

SUMMARY:
To evaluate the safety and tolerability of Nitazoxanide (NTZ) 500mg Twice Daily (BID) after 24 weeks of treatment in patients with NASH induced Stage 2 or Stage 3 fibrosis

DETAILED DESCRIPTION:
Based on the anti-fibrotic properties demonstrated in the animal models of fibrosis, this proof of concept clinical study aims at evaluating NTZ in patients with non-alcoholic steatohepatitis (NASH) and fibrosis stage 2 and 3. Although NTZ has been evaluated in liver disease populations up to 60 weeks, this is the first study evaluating NTZ treatment in a population with NASH induced stage 2 and 3 fibrosis. The aim of this study is to evaluate the safety and tolerability of NTZ 500 mg BID after 24 weeks of treatment in this population.

This proof of concept study will also evaluate the anti-fibrotic effect of NTZ as a secondary objective.

The methods of evaluation of fibrosis will include an innovative method of metabolic labeling.This approach is based on the concept that liver status can be determined by measuring the ratio of newly synthesized/pre-existing proteins.The turn-over rate of newly synthesized collagen and proteins represents the hepatic fibrogenic disease activity. Patients will be given "heavy water" to drink. Heavy water contains D20, deuterium being a stable isotope of hydrogen. Mass spectrometry is used to identify individual proteins and to quantify the ratio of labeled protein to total protein. The results are expressed as fractional synthesis rate of these proteins (FSR). This method has been previously published (Decaris et al, 2017).

Other non-invasive methods will be used to evaluate the liver stiffness changes after NTZ treatment: Magnetic Resonance Elastography (MRE) and FibroScan®.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged from 18 to 75 years inclusive the Screening Visit.
2. Must provide signed written informed consent and agree to comply with the study protocol.
3. Females participating in this study must be of non-childbearing potential or using highly efficient contraception for the full duration of the study
4. Histological confirmation of steatohepatitis on a diagnostic liver biopsy (biopsy obtained within 6 months prior to Screening or during the Screening Period) with at least 1 in each component of the NAS (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3).
5. Fibrosis stage of 2 or 3, according to the NASH Clinical Research Network fibrosis staging system on a diagnostic liver biopsy (biopsy obtained within 6 months prior to Screening or during the Screening Period).
6. Two assessments of ALT, AST, Total bilirubin, Alkaline phosphatase (ALP), Creatine phosphokinase (CPK) will be collected during screening at least 4 weeks apart. To be eligible the second value cannot be ≥2x the first value.

Exclusion Criteria:

1. History of efficient bariatric surgery within 5 years prior to Screening, or planned bariatric surgery in the course of the study.
2. Patients with HbA1c >10.0%. If abnormal at the first Screening Visit, the HbA1c measurement can be repeated. A repeated abnormal HbA1c (HbA1c >10.0%) leads to exclusion.
3. Patients with a history of clinically significant acute cardiac event within 6 months prior to Screening such as: stroke, transient ischemic attack, or coronary heart disease (angina pectoris, myocardial infarction, revascularization procedures).
4. Weight loss of more than 10% within 6 months prior to Randomization.
5. Patient with any history or presence of decompensated cirrhosis.
6. Current or recent history (<1 year) of significant alcohol consumption. For men, significant consumption is typically defined as higher than 30 g pure alcohol per day. For women, it is typically defined as higher than 20 g pure alcohol per day.
7. Current or history of other substance abuse within 1 year prior to screening.
8. Pregnant or lactating females or females planning to become pregnant during the study period.
9. Other well documented causes of chronic liver disease according to standard diagnostic procedures including, but not restricted to:

   1. Positive hepatitis B surface antigen (HBsAg)
   2. Positive Hepatitis C virus (HCV) RNA, (tested for in case of known cured HCV infection, or positive HCV Ab at Screening)
   3. Suspicion of drug-induced liver disease
   4. Alcoholic liver disease
   5. Autoimmune hepatitis
   6. Wilson's disease
   7. Primary biliary cirrhosis, primary sclerosing cholangitis
   8. Genetic homozygous hemochromatosis
   9. Known or suspected Hepatocellular Carcinoma
   10. History or planned liver transplant, or current Model for End-Stage Liver Disease score >15.
10. Patients who cannot be contacted in case of emergency.
11. Known hypersensitivity to the investigation product or any of its formulation excipients.
12. Patients who are taking warfarin or other highly plasma protein-bound drugs with narrow therapeutic indices.
13. Patients who are currently participating in, plan to participate in, or have participated in an investigational drug trial or medical device trial containing active substance within 30 days or five half-lives, whichever is longer, prior to Screening.
14. Evidence of any other unstable or, untreated clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic, or psychiatric disease.
15. Mental instability or incompetence, such that the validity of informed consent or ability to be compliant with the study is uncertain.
16. History of noncompliance with medical regimens, or patients who are considered to be unreliable.
17. Positive anti-human immunodeficiency virus (HIV) antibody.
18. AST and/or ALT >10 x upper limit of normal (ULN).
19. Total bilirubin >1.3 mg/dL due to altered hepatic function.
20. Direct bilirubin > ULN Note: Gilbert Disease patients are allowed into the study.
21. International Normalized Ratio >1.2 in the absence of anticoagulant therapy.
22. Platelet count <150,000/mm3 in the context of portal hypertension.
23. Significant renal disease, including nephritic syndrome, chronic kidney disease (defined as patients with markers of kidney damage or estimated glomerular filtration rate of less than 60 ml/min/1.73 m2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Pinnacle Clinical Research
Locations (1):
- Pinnacle Clinical Research, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female patients aged from 18 to 75 years, inclusive, at the Screening Visit, with histologically confirmed NASH and fibrosis Stage 2 or 3 were enrolled in the study at a single research center in the United States, at Pinnacle Clinical Research, 5109 Medical Drive, Suite 200 San Antonio, TX 78229.
Pre-assignment Details: Potential Subjects who completed all of the Screening Visit assessments and who continued to be eligible for the study, returned to the research center to complete a deuterated water Run-In period. The visit was done on Day -14 +/- 3 days, provided that the subject completed 7 consecutive days of deuterated water administration. Patients returned at Day-11, Day-7 (+/- 1 day) and Day 1 for blood sampling (labelled D2O).
Groups:
- NTZ 500 mg BID: Open label group: all patients were to receive study drug Nitazoxanide (Alinia) 500 mg BID for 24 weeks.
Period: Overall Study
Arm/Group | NTZ 500 mg BID
Started | 21
Completed | 16
Not Completed | 5
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- NTZ 500 mg BID: Open label group: all patients were to receive study drug Nitazoxanide 500mg BID for 24 weeks.
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Height at Screening [Mean (Standard Deviation); unit: cm] | 164.4 (9.17)
Baseline weight [Mean (Standard Deviation); unit: kg] | 94.14 (17.793)
Baseline body mass index [Mean (Standard Deviation); unit: kg/m²] | 34.64 (4.638)

OUTCOME MEASURES:

1. Primary Outcome: Number of NTZ Treated Participants Presenting Any Treatment Emergent Adverse Event (TEAE)
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of treatment-emergent adverse events (TEAEs).
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  No of participants with at least one TEAE | 20
  TEAE maximum severity: Grade 1 (mild) | 7
  TEAE maximum severity: Grade 2 (moderate) | 10
  TEAE maximum severity: Grade 3 (severe) | 3
  TEAE maximum severity: Grade 4 (life-threatening) | 0
  TEAE maximum severity: Grade 5 (death) | 0
  No of participants with no TEAE | 1

2. Primary Outcome: Number of NTZ Treated Participants Presenting Any Study Drug Related TEAE
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of study drug-related treatment-emergent adverse events (TEAEs).
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  No of participants with at least 1 treatment-related TEAE | 18
  TEAE maximum severity: Grade 1 (mild) | 10
  TEAE maximum severity: Grade 2 (moderate) | 8
  TEAE maximum severity: Grade 3 (severe) | 0
  TEAE maximum severity: Grade 4 (life-threatening) | 0
  TEAE maximum severity: Grade 5 (death) | 0
  No of participants with no study drug-related TEAE | 3

3. Primary Outcome: Number of NTZ Treated Participants Presenting Any SAE
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of serious adverse events (SAEs).
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one SAE | 4
  No SAE | 17

4. Primary Outcome: Number of NTZ Treated Participants Presenting Study Drug-Related SAE
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of study drug-related serious adverse events (SAEs).
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one study-drug related SAE | 0
  No study-drug related SAE | 21

5. Primary Outcome: Deaths Due to AE
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of deaths due to adverse events (AEs).
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  Yes | 0
  No | 21

6. Primary Outcome: Number of NTZ Treated Participants Presenting Any AE Leading to Withdrawal From Study or Study Drug
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of adverse events (AEs) leading to withdrawal from study or study drug.
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one AE leading to withdrawal | 1
  No AE leading to withdrawal | 20

7. Primary Outcome: Number of NTZ Treated Participants Presenting Any Study Drug-related AE Leading to Withdrawal From Study or Study Drug
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by assessing the occurrence of study drug-related adverse events (AEs) leading to withdrawal from study or study drug
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one study drug-related AE leading to withdrawal | 0
  No study drug-related AE leading to withdrawal | 21

8. Primary Outcome: Number of NTZ Treated Participants Presenting at Least One Clinically Significant (CS) Change in Clinical Laboratory Evaluations
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by performing clinical laboratory evaluations. Changes in clinical laboratory evaluations were considered clinically significant or not as per Investigator judgment.
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one CS change | 0
  No CS change | 21

9. Primary Outcome: Number of NTZ Treated Participants Presenting at Least One Clinically Significant (CS) Change in Vital Signs
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by measuring vital signs. Changes in vital signs were considered clinically significant or not as per Investigator judgement
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one CS change | 0
  No CS change | 21

10. Primary Outcome: Number of NTZ Treated Participants Presenting at Least One Clinically Significant (CS) Change in Electrocardiogram Parameters
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by performing electrocardiograms (ECGs). Changes in ECGs parameters were considered clinically significant or not as per Investigator judgement.
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one CS change | 0
  No CS change | 21

11. Primary Outcome: Number of NTZ Treated Participants Presenting at Least One Clinically Significant (CS) Change in Physical Examinations
Description: To assess the safety and tolerability of NTZ after 24 weeks of treatment by conducting physical examinations. Changes in physical examinations were considered clinically significant or not as per Investigator judgement.
Time Frame: 28 weeks
Population: The Safety Analysis Set consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
Participants
  At least one CS change | 0
  No CS change | 21

12. Secondary Outcome: Change in Lumican Fractional Synthesis Rate (FSR) From Baseline to End of Treatment
Description: Change in Lumican Fractional Synthesis Rate (FSR) from baseline to end of treatment evaluated through the use of deuterated water.
  Lumican is a marker indicative of hepatic fibrogenesis with its turnover assessed by Fractional Synthesis Rate (FSR). This innovative method of metabolic labelling is based on the concept that liver status could be determined by measuring the ratio of newly synthesized/pre-existing proteins. The turnover rate of newly synthesized collagen and proteins represents the hepatic fibrogenic disease activity.
  Patients were given "heavy water" to drink. Heavy water contains D20, deuterium being a stable isotope of hydrogen. Mass spectrometry was used to identify individual proteins and to quantify the ratio of labeled protein to total protein.
Time Frame: From baseline to end of treatment (Visit 10, Week 24 or early termination)
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
Measure: Mean (Standard Deviation); unit: pools per day
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
pools per day | 0.0046 (0.00924)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Wilcoxon signed-rank test was used for statistical inference; p = 0.0039, Sign test — p-value for testing median = 0; Median Difference (Net) = 0.0030

13. Secondary Outcome: Percent Change in Lumican Fractional Synthesis Rate (FSR) From Baseline to End of Treatment
Description: Percent Change in Lumican FSR from baseline to end of treatment evaluated through the use of deuterated water.
  Lumican is a marker indicative of hepatic fibrogenesis with its turnover assessed by Fractional Synthesis Rate (FSR). This innovative method of metabolic labelling is based on the concept that liver status could be determined by measuring the ratio of newly synthesized/pre-existing proteins. The turnover rate of newly synthesized collagen and proteins represents the hepatic fibrogenic disease activity.
  Patients were given "heavy water" to drink. Heavy water contains D20, deuterium being a stable isotope of hydrogen. Mass spectrometry was used to identify individual proteins and to quantify the ratio of labeled protein to total protein.
Time Frame: From baseline to end of treatment (Visit 10, Week 24 or early termination)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 15.46 (22.507)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Wilcoxon signed-rank test was used for statistical inference; p = 0.0026, Sign test — p-value for testing median = 0; Median Difference (Net) = 10.00

14. Secondary Outcome: Change in Transforming Growth Factor Beta-induced Protein (TGFBI) FSR From Baseline to End of Treatment
Description: Change in transforming growth factor beta-induced-protein (TGFBI) Fractional Synthesis Rate (FSR) from baseline to end of treatment evaluated through the use of deuterated water.
  TGFBI is a marker indicative of hepatic fibrogenesis with its turnover assessed by FSR.
  This innovative method of metabolic labelling is based on the concept that liver status could be determined by measuring the ratio of newly synthesized/pre-existing proteins. The turnover rate of newly synthesized collagen and proteins represents the hepatic fibrogenic disease activity.
  Patients were given "heavy water" to drink. Heavy water contains D20, deuterium being a stable isotope of hydrogen. Mass spectrometry was used to identify individual proteins and to quantify the ratio of labeled protein to total protein. The results were expressed as FSR of these proteins.
Time Frame: From baseline to end of treatment (Visit 10, Week 24 or early termination)
Measure: Mean (Standard Deviation); unit: pools per day
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
pools per day | 0.0014 (0.01124)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Wilcoxon signed-rank test was used for statistical inference; p = 0.5555, Sign test — p-value for testing median = 0; Median Difference (Net) = 0.0020

15. Secondary Outcome: Percent Change in Transforming Growth Factor Beta-induced Protein (TGFBI) FSR From Baseline to End of Treatment
Description: Percent Change in transforming growth factor beta-induced protein (TGFBI) FSR from baseline to end of treatment evaluated through the use of deuterated water.
  TGFBI is a marker indicative of hepatic fibrogenesis with its turnover assessed by Fractional Synthesis Rate (FSR).
  This innovative method of metabolic labelling is based on the concept that liver status could be determined by measuring the ratio of newly synthesized/pre-existing proteins. The turnover rate of newly synthesized collagen and proteins represents the hepatic fibrogenic disease activity.
  Patients were given "heavy water" to drink. Heavy water contains D20, deuterium being a stable isotope of hydrogen. Mass spectrometry was used to identify individual proteins and to quantify the ratio of labeled protein to total protein. The results were expressed as FSR of these proteins.
Time Frame: From baseline to end of treatment (Visit 10, Week 24 or early termination)
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 3.20 (12.619)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Wilcoxon signed-rank test was used for statistical inference; p = 0.3778, Sign test — p-value for testing median = 0; Median Difference (Net) = 1.72

16. Secondary Outcome: Change in Controlled Attenuation Parameter (CAP) Score From Baseline to End of Treatment as Evaluated by FibroScan®
Description: FibroScan is a specialized ultrasound machine that measures fibrosis (scarring) and steatosis (fatty change) in the liver. It was required that each subject's FibroScan® assessments be done with the same type of probe at each study visit.
  The CAP score is a measurement of fatty change in the liver, naming the steatosis grade. The CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m. 100 to 237 dB/M indicates no hepatic steatosis, 238 to 260 dB/m indicates mild hepatic steatosis (steatosis S1), 260 to 290 dB/m indicates moderate steatosis (steatosis S2), and a CAP score greater than 290 dB/m indicates severe steatosis (steatosis S3).
Time Frame: 24 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: dB/m
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
dB/m | -8.1 (44.59)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.4638, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -8.1, 95% CI 2-sided [-31.0 to 14.8]

17. Secondary Outcome: Percent Change in Controlled Attenuation Parameter (CAP) Score From Baseline to End of Treatment as Evaluated by FibroScan®
Description: FibroScan is a specialized ultrasound machine that measures fibrosis (scarring) and steatosis (fatty change) in the liver. It was required that each subject's FibroScan® assessments be done with the same type of probe at each study visit.
  The CAP score is a measurement of fatty change in the liver, naming the steatosis grade.The CAP score is measured in decibels per meter (dB/m). It ranges from 100 to 400 dB/m. 100 to 237 dB/M indicates no hepatic steatosis, 238 to 260 dB/m indicates mild hepatic steatosis (steatosis S1), 260 to 290 dB/m indicates moderate steatosis (steatosis S2), and a CAP score greater than 290 dB/m indicates severe steatosis (steatosis S3).
Time Frame: 24 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -1.65 (14.818)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.6532, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -1.65, 95% CI 2-sided [-9.26 to 5.97]

18. Secondary Outcome: Change in Liver Stiffness From Baseline to End of Treatment as Evaluated by FibroScan®
Description: FibroScan is a specialized ultrasound machine that measures fibrosis (scarring) and steatosis (fatty change) in the liver. It was required that each subject's FibroScan® assessments be done with the same type of probe at each study visit.
  The fibrosis result is measured in kilopascals (kPa) It's normally between 2 and 6 kPa indicating the abscence of abscence of fibrosis (F0) or a potential fibrosis of stage 1 (F1). The highest possible result is 75 kPa indicating advanced liver fibrosis of stage 4 (F4).
Time Frame: 24 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
kPa | 0.38 (4.341)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7254, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.38, 95% CI 2-sided [-1.86 to 2.61]

19. Secondary Outcome: Percent Change in Liver Stiffness From Baseline to End of Treatment as Evaluated by FibroScan®
Description: as for outcome 18
Time Frame: 24 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 8.77 (39.828)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3772, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 8.77, 95% CI 2-sided [-11.70 to 29.25]

20. Secondary Outcome: Change in Liver Stiffness From Baseline to Week 12 as Evaluated Through the Use Magnetic Resonance Elastography (MRE)
Description: Liver stiffness was assessed by MRE. It was recommended that each subject's radiological assessment was performed using the same procedure for each study visit.
Time Frame: 12 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 13 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the week 12 visit.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 13
kPa | -0.12 (0.731)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.5799, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.56 to 0.33]

21. Secondary Outcome: Percent Change in Liver Stiffness From Baseline to Week 12 as Evaluated Through the Use Magnetic Resonance Elastography (MRE)
Description: as for outcome 20
Time Frame: 12 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 13
percentage of change | -1.89 (17.807)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7088, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -1.89, 95% CI 2-sided [-12.65 to 8.87]

22. Secondary Outcome: Change in Liver Stiffness From Baseline to End of Treatment as Evaluated Through the Use Magnetic Resonance Elastography (MRE)
Description: as for outcome 20
Time Frame: 24 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 12 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the end of treatment visit.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 12
kPa | -0.35 (0.581)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0609, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.72 to 0.02]

23. Secondary Outcome: Percent Change in Liver Stiffness From Baseline to End of Treatment as Evaluated Through the Use Magnetic Resonance Elastography (MRE)
Description: as for outcome 20
Time Frame: 24 weeks
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 12
percentage of change | -6.61 (15.029)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1556, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -6.61, 95% CI 2-sided [-16.16 to 2.94]

24. Secondary Outcome: Change in Alpha-2 Macroglobulin From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  21 patients were analyzed for this Outcome Measure, as all patients had a result both at baseline and at the week 12 visit.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
mg/dL | -11.0 [-94 to 56]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0709, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -14.6, 95% CI 2-sided [-30.6 to 1.4]

25. Secondary Outcome: Percent Change in Alpha-2 Macroglobulin From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | -5.64 [-20.0 to 27.3]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1799, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -3.61, 95% CI 2-sided [-9.02 to 1.81]

26. Secondary Outcome: Change in Alpha-2 Macroglobulin From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 17 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the end of treatment visit.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
mg/dL | -9.0 [-70 to 42]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3306, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -6.8, 95% CI 2-sided [-21.2 to 7.6]

27. Secondary Outcome: Percent Change in Alpha-2 Macroglobulin From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -4.85 [-16.0 to 22.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.4504, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -1.94, 95% CI 2-sided [-7.25 to 3.37]

28. Secondary Outcome: Change in Fibroblast Growth Factor 19 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 20 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the week 12 visit.
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
ng/L | 28.0 [-155 to 282]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1349, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 33.8, 95% CI 2-sided [-11.5 to 79.0]

29. Secondary Outcome: Percent Change in Fibroblast Growth Factor 19 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
percentage of change | 38.74 [-68.9 to 361.1]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0117, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 76.24, 95% CI 2-sided [19.04 to 133.43]

30. Secondary Outcome: Change in Fibroblast Growth Factor 19 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
ng/L | 24.0 [-377 to 290]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.4281, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 31.3, 95% CI 2-sided [-50.3 to 112.9]

31. Secondary Outcome: Percent Change in Fibroblast Growth Factor 19 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 42.11 [-81.1 to 637.8]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0407, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 117.37, 95% CI 2-sided [5.60 to 229.14]

32. Secondary Outcome: Change in Fibroblast Growth Factor 21 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
ng/L | 2.40 [-1609.8 to 1009.8]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7065, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 47.28, 95% CI 2-sided [-210.90 to 305.46]

33. Secondary Outcome: Percent Change in Fibroblast Growth Factor 21 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | 0.36 [-68.6 to 504.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1693, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 43.11, 95% CI 2-sided [-19.95 to 106.17]

34. Secondary Outcome: Change in Fibroblast Growth Factor 21 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
ng/L | -102.90 [-1728.6 to 928.9]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7099, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -48.14, 95% CI 2-sided [-317.64 to 221.36]

35. Secondary Outcome: Percent Change in Fibroblast Growth Factor 21 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -15.36 [-56.8 to 511.8]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3597, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 30.03, 95% CI 2-sided [-37.48 to 97.55]

36. Secondary Outcome: Change in Human Chitinase 3-like 1 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
ng/L | 5423.0 [-180529 to 91341]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9893, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 169.0, 95% CI 2-sided [-25908.2 to 26246.2]

37. Secondary Outcome: Percent Change in Human Chitinase 3-like 1 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | 8.90 [-54.0 to 106.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1454, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 13.82, 95% CI 2-sided [-5.21 to 32.85]

38. Secondary Outcome: Change in Human Chitinase 3-like 1 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: ng/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
ng/L | 5338.0 [-102066 to 121135]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.8089, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 3016.8, 95% CI 2-sided [-22996.2 to 29029.7]

39. Secondary Outcome: Percent Change in Human Chitinase 3-like 1 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 8.76 [-36.8 to 74.9]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1365, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 12.78, 95% CI 2-sided [-4.50 to 30.06]

40. Secondary Outcome: Change in Hyaluronic Acid From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
µg/L | 6.210 [-22.12 to 323.24]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1322, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 28.954, 95% CI 2-sided [-9.525 to 67.433]

41. Secondary Outcome: Percent Change in Hyaluronic Acid From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | 10.93 [-41.1 to 199.3]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1062, t-test, 2 sided; p-value for testing mean = 0; Mean Difference (Net) = 23.99, 95% CI 2-sided [-5.59 to 53.57]

42. Secondary Outcome: Change in Hyaluronic Acid From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
µg/L | 6.100 [-26.83 to 235.19]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0831, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 28.311, 95% CI 2-sided [-4.151 to 60.774]

43. Secondary Outcome: Percent Change in Hyaluronic Acid From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 6.99 [-46.2 to 202.2]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0543, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 32.72, 95% CI 2-sided [-0.69 to 66.13]

44. Secondary Outcome: Change in Liver Fibrosis Score Enhanced Liver Fibrosis (ELF) From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples. ELF score is a continuous (not a categorical) variable with < 9.8 indicative of low risk of progression to cirrhosis and >=9.8 to >11.3 indicative of mid-risk and >=11.30 indicative of higher risk
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
score | -0.160 [-0.67 to 1.25]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.6325, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.056, 95% CI 2-sided [-0.185 to 0.298]

45. Secondary Outcome: Percent Change in Liver Fibrosis Score Enhanced Liver Fibrosis (ELF) From Baseline to Week 12
Description: as for outcome 44
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | -1.64 [-7.3 to 11.5]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.6925, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.46, 95% CI 2-sided [-1.94 to 2.87]

46. Secondary Outcome: Change in Liver Fibrosis Score Enhanced Liver Fibrosis (ELF) From Baseline to End of Treatment
Description: as for outcome 44
Time Frame: 24 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 16 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the end of treatment visit.
Measure: Median (Full Range); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
score | 0.090 [-0.89 to 1.32]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.2733, t-test, 2 sided; Mean Difference (Net) = 0.161, 95% CI 2-sided [-0.140 to 0.462]

47. Secondary Outcome: Percent Change in Liver Fibrosis Score Enhanced Liver Fibrosis (ELF) From Baseline to End of Treatment
Description: as for outcome 44
Time Frame: 24 weeks
Population: as for outcome 46
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
percentage of change | 0.90 [-9.7 to 12.0]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3288, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 1.47, 95% CI 2-sided [-1.63 to 4.56]

48. Secondary Outcome: Change in M30 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Median (Full Range); unit: U/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
U/L | 0.000 [-500.92 to 740.29]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9271, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 5.649, 95% CI 2-sided [-121.923 to 133.220]

49. Secondary Outcome: Percent Change in M30 Biomarker From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
percentage of change | 0.00 [-59.7 to 89.2]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9244, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.89, 95% CI 2-sided [-18.58 to 20.37]

50. Secondary Outcome: Change in M30 Biomarker From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: U/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
U/L | -34.920 [-602.50 to 853.74]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7288, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -30.244, 95% CI 2-sided [-211.930 to 151.441]

51. Secondary Outcome: Percent Change in M30 Biomarker From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -5.48 [-63.9 to 113.0]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7824, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 3.34, 95% CI 2-sided [-21.85 to 28.52]

52. Secondary Outcome: Change in M65 Biomarker From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Median (Full Range); unit: U/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
U/L | -15.605 [-1100.35 to 801.43]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.6448, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -47.629, 95% CI 2-sided [-260.433 to 165.176]

53. Secondary Outcome: Percent Change in M65 Biomarker From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
percentage of change | -3.52 [-90.7 to 144.2]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9806, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.38, 95% CI 2-sided [-32.04 to 32.80]

54. Secondary Outcome: Change in M65 Biomarker From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: U/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
U/L | -58.970 [-1098.60 to 839.44]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3256, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -113.616, 95% CI 2-sided [-351.124 to 123.891]

55. Secondary Outcome: Percent Change in M65 Biomarker From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -11.56 [-84.6 to 213.2]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.6582, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 8.78, 95% CI 2-sided [-32.52 to 50.09]

56. Secondary Outcome: Change in miR34a Fold From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 16 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the week 12 visit.
Measure: Median (Full Range); unit: fold change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
fold change | -0.0991 [-4.331 to 2.033]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.5459, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.2438, 95% CI 2-sided [-1.0847 to 0.5972]

57. Secondary Outcome: Percent Change in miR34a Fold From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 56
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
percentage of change | -7.42 [-66.3 to 213.8]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.2860, t-test, 2 sided; Mean Difference (Net) = 23.91, 95% CI 2-sided [-22.15 to 69.97]

58. Secondary Outcome: Change in miR34a Fold From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 46
Measure: Median (Full Range); unit: fold change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
fold change | -0.5019 [-3.561 to 3.181]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.4887, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.2893, 95% CI 2-sided [-1.1580 to 0.5794]

59. Secondary Outcome: Percent Change in miR34a Fold From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 46
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 16
percentage of change | -24.90 [-78.1 to 308.4]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3610, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 30.27, 95% CI 2-sided [-38.21 to 98.75]

60. Secondary Outcome: Change in Pro-C3 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
µg/L | -0.80 [-8.0 to 10.8]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.4945, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.63, 95% CI 2-sided [-2.51 to 1.26]

61. Secondary Outcome: Percent Change in Pro-C3 From Baseline to Week 12
Description: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | -2.80 [-28.7 to 59.3]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.8191, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.99, 95% CI 2-sided [-9.94 to 7.95]

62. Secondary Outcome: Change in Pro-C3 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
µg/L | -2.60 [-14.8 to 6.3]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0243, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -3.22, 95% CI 2-sided [-5.96 to -0.47]

63. Secondary Outcome: Percent Change in Pro-C3 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -12.70 [-42.5 to 34.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0493, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -9.94, 95% CI 2-sided [-19.84 to -0.04]

64. Secondary Outcome: Change in Pro-C6 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
µg/L | 0.40 [-2.6 to 9.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3066, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.60, 95% CI 2-sided [-0.59 to 1.79]

65. Secondary Outcome: Percent Change in Pro-C6 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | 1.98 [-14.4 to 36.2]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.2671, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 3.40, 95% CI 2-sided [-2.82 to 9.63]

66. Secondary Outcome: Change in Pro-C6 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
µg/L | -0.20 [-4.4 to 3.9]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.8241, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.94 to 1.16]

67. Secondary Outcome: Percent Change in Pro-C6 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | -0.75 [-24.3 to 24.5]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.7587, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 1.10, 95% CI 2-sided [-6.37 to 8.57]

68. Secondary Outcome: Change in Procollagen 3 N-terminal Pro-peptide From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
µg/L | -1.560 [-4.46 to 5.38]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3784, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.567, 95% CI 2-sided [-1.880 to 0.746]

69. Secondary Outcome: Percent Change in Procollagen 3 N-terminal Pro-peptide From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | -9.73 [-33.5 to 34.9]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3526, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -4.64, 95% CI 2-sided [-14.80 to 5.53]

70. Secondary Outcome: Change in Procollagen 3 N-terminal Pro-peptide From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
µg/L | 0.180 [-5.22 to 11.83]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9218, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.098, 95% CI 2-sided [-1.978 to 2.173]

71. Secondary Outcome: Percent Change in Procollagen 3 N-terminal Pro-peptide From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 1.22 [-42.9 to 59.1]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.9833, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 0.15, 95% CI 2-sided [-14.71 to 15.01]

72. Secondary Outcome: Change in Tissue Inhibitor of Metalloproteinase 1 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
µg/L | 10.50 [-133.2 to 177.5]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3957, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 12.68, 95% CI 2-sided [-17.79 to 43.16]

73. Secondary Outcome: Percent Change in Tissue Inhibitor of Metalloproteinase 1 From Baseline to Week 12
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 12 weeks
Population: as for outcome 24
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 21
percentage of change | 3.53 [-21.1 to 38.0]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3440, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 3.81, 95% CI 2-sided [-4.39 to 12.01]

74. Secondary Outcome: Change in Tissue Inhibitor of Metalloproteinase 1 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: µg/L
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
µg/L | 13.40 [-36.6 to 67.4]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0607, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 15.22, 95% CI 2-sided [-0.77 to 31.21]

75. Secondary Outcome: Percent Change in Tissue Inhibitor of Metalloproteinase 1 From Baseline to End of Treatment
Description: Non-invasive Fibrosis Biomarkers were assessed in blood samples.
Time Frame: 24 weeks
Population: as for outcome 26
Measure: Median (Full Range); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 17
percentage of change | 3.78 [-16.6 to 27.6]
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0644, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 5.83, 95% CI 2-sided [-0.39 to 12.05]

76. Secondary Outcome: Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score From Baseline to Week 12
Description: NAFLD NFS : < -1.5 for low probability of fibrosis, > -1.5 to < 0.67 for intermediate probability of fibrosis, and > 0.67 for high probability of fibrosis.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
score | -0.3665 (0.77812)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.0487, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.3665, 95% CI 2-sided [-0.7306 to -0.0023]

77. Secondary Outcome: Percent Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score From Baseline to Week 12
Description: as for outcome 76
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
percentage of change | 16.64 (136.529)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.5919, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 16.64, 95% CI 2-sided [-47.25 to 80.54]

78. Secondary Outcome: Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score From Baseline to End of Treatment
Description: as for outcome 76
Time Frame: 24 weeks
Population: The Full Analysis Set consisted of all patients who met the eligibility criteria and enrolled into the study (Visit 1 Day 1).
  There were 8 patients analyzed for this Outcome Measure, corresponding to the patients having a result both at baseline and at the end of treatment visit.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 8
score | -0.2679 (0.43795)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1272, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.2679, 95% CI 2-sided [-0.6340 to 0.0983]

79. Secondary Outcome: Percent Change in Non-Alcoholic Fatty Liver Disease (NAFLD) Fibrosis Score From Baseline to End of Treatment
Description: as for outcome 76
Time Frame: 24 weeks
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 8
percentage of change | 15.02 (74.847)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.5881, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = 15.02, 95% CI 2-sided [-47.55 to 77.59]

80. Secondary Outcome: Change in Fibrosis-4 Score From Baseline to Week 12
Description: Fibrosis-4 score : FIB4 < 1.3 is not consistent with F3-F6 disease. FIB4 of 1.3 to <2.67 is indeterminate for F3-F6 disease. > 2.67 is consistent F3 to F6.
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
score | -0.18 (0.516)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1458, t-test, 2 sided; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.42 to 0.07]

81. Secondary Outcome: Percent Change in Fibrosis-4 Score From Baseline to Week 12
Description: as for outcome 80
Time Frame: 12 weeks
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 20
percentage of change | -11.53 (34.342)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.1495, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -11.53, 95% CI 2-sided [-27.61 to 4.54]

82. Secondary Outcome: Change in Fibrosis-4 Score From Baseline to End of Treatment
Description: as for outcome 80
Time Frame: 24 weeks
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: score
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 8
score | -0.12 (0.328)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.3174, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.40 to 0.15]

83. Secondary Outcome: Percent Change in Fibrosis-4 Score From Baseline to End of Treatment
Description: as for outcome 80
Time Frame: 24 weeks
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | NTZ 500 mg BID
Number analyzed (Participants) | 8
percentage of change | -8.02 (17.754)
Statistical Analysis 1: Comparison: NTZ 500 mg BID; Test type: Other — Student's T-test was used for statistical inference; p = 0.2420, t-test, 2 sided — p-value for testing mean = 0; Mean Difference (Net) = -8.02, 95% CI 2-sided [-22.86 to 6.82]

ADVERSE EVENTS:
Time Frame: from the signature of the informed consent form (ICF) until the end of study, week 28, i.e. 4 weeks after the last administration.
Description: All AEs regardless of seriousness or relationship to study drug, including those occurring during the Screening Period, were recorded in the eCRF from ICF signature until study end for each patient. Whenever possible, symptoms were grouped as a single syndrome or diagnosis.
  The Investigator established whether or not any AE occurred at each visit from the date of consent. The patient was questioned in a general manner without offering the patient any suggestion.
Arm/Group | NTZ 500 mg BID
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTZ 500 mg BID (N=21)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) — worsening of symptomatic menometrorrhagia
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Paroxysmal atrial fibrillation with rapid ventricular response
Angina Unstable (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) — worsening of coronary artery disease
cardiac failure (Cardiac disorders) | 1 (1) — worsening of heart failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NTZ 500 mg BID (N=21)
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pancreatic cyst (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Chromaturia (Renal and urinary disorders) | 7
Ureterolithiasis (Renal and urinary disorders) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Glomerular filtration rate increased (Investigations) | 1
Glycosylated haemoglobin increased (Investigations) | 1
Heart rate increased (Investigations) | 1
Norovirus test positive (Investigations) | 1
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Hypertryglyceridaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
fall (Injury, poisoning and procedural complications) | 3
Arthropod sting (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 2
Fatigue (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Vision blurred (Eye disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (8):
  • Study Protocol: V27AUG2018 (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_000.pdf
  • Study Protocol: V21OCT2018 (2018-10-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_001.pdf
  • Study Protocol: V02MAR2019 (2019-03-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_002.pdf
  • Study Protocol: V24AUG2019 (2019-08-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_003.pdf
  • Study Protocol: 26FEB2020 (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_004.pdf
  • Study Protocol: V15APR2020 (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/Prot_005.pdf
  • Statistical Analysis Plan: V1.0 (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/SAP_006.pdf
  • Statistical Analysis Plan: V1.1 (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03656068/SAP_007.pdf